CLINICAL TRIAL: NCT04728490
Title: Haplo-identical Transplantation in Patients With Myelofibrosis - A Phase 2 Prospective Multicentric Prospective Study
Acronym: FIBRAPLO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP190648
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogenic transplantation using treosulfan in conditioning regimen (Experimental): Haplo-identical transplantation using treosulfan in conditioning regimen Treosuflan, in the conditioning regimen will be administrated as followed 10 gr/m2 per day -4, -3 and -2 IV route
  In combination with:
  Thiotepa 5 mg/kg on day -6 Fludarabine 30 mg/m2 per day from day -5 to day -1
  Interventions: Other: Allogenic transplantation transplantation

INTERVENTIONS:
Other: Allogenic transplantation transplantation — Haplo-identical transplantation with the use of Treosulfan, Thiotepa and Fludarabine in conditioning regimen.

SUMMARY:
The only curative treatment in patients with primary or secondary myelofibrosis is allogeneic hematopoietic stem cells (HSCT). It has been reported that intermediate and higher risk patients according to international prognostic scores benefit from HSCT in terms of survival (Kröger et al, 2015). In 2013, we conducted in France a prospective trial testing the use of ruxolitinib before transplantation ("JAK-ALLO study" NCT01795677). Outcome of patients was better in patients transplanted with a matched sibling donor than an unrelated donor confirming other studies (Kröger et al, 2009; Rondelli et al, 2014). In the JAK-ALLO trial, acute GVHD incidence was high, often hyperacute and severe. Recently, the EBMT group has reported a registry study on familial haplo-identical transplantation (haplo) in patients with myelofibrosis (Raj et al, 2018). Post-transplant cyclophosphamide was used in 59% of cases. One-year overall survival (OS) and disease-free survival (DFS) were 61 and 58% which favorably compared to outcome after unrelated transplantation. Genova team has also reported impressive results after haplo-identical transplantation in their center (Bregante et al, 2015). Bregante et al have reported outcome of 2 cohorts transplanted from 2000 to 2010 and from 2011 to 2014. The main difference between the 2 periods is the more frequent use of haplo in the second period (54% versus 5%). Outcome was much better in the second period with OS at 70% versus 49% and authors suggest that this improvement is related to the best outcome among haplo transplantation. The improvement of outcome after haplo has been attributed to a better GVHD prophylaxis, especially with the use of post-transplant cyclophosphamide. Given the poor outcome after unrelated transplantation and especially in HLA mismatched unrelated setting and encouraging results in family haplo identical transplantation, this current study proposes to test haplo-identical transplantation in myelofibrosis patients without a matched related donor.

The main objective of this study is disease and rejection-free survival one year after haplo-identical transplantation in patients with primary or secondary myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years
* Primary myelofibrosis or myelofibrosis secondary to essential thrombocythemia or polycythemia Vera proven by marrow biopsy
* The myelofibrosis should combine at least 2 of the following criteria:

  * constitutional symptoms: weight loss > 10% in one year, fever (without infection), recurrent muscle, bone or join pains, extreme fatigue
  * anemia with hemoglobin < 10 gr/dL or red blood cell transfusion requirement
  * thrombocytopenia < 100 G/L
  * peripheral blast count > 1% at least found 2 times
  * white blood cell count > 25 G/L (before a cytoreductive treatment)
  * Karyotype: +8, -7/7q-, i(17q), -5, 5q-, 12p-, inv(3), 11q23
* Performance status according to ECOG at 0, 1 or 2
* With health insurance coverage
* Having signed a written informed consent
* Women agreed to take nomegestrol acetate as contraception during and up to 6 months after treatment by treosulfan
* Men agreed not to conceive child during and up to 6 months after treatment by treosulfan

Exclusion Criteria:

* Myelofibrosis transformed into acute leukemia
* Poor performance status with ECOG 3 or more
* Cardiac failure with EF < or = 50% currently or in the past (even if corrected after treatment)
* Renal failure with creatininemia > 130 µmol/L or clearance < 50ml/min
* Respiratory function altered with vital capacity < 70% or forced expired volume < 70%
* Biological significant liver abnormalities; ASAT or ALAT> 2 x normal range, bilirubin > 1,5 x normal range
* HLA matched donor available
* Tutorship or curatorship
* Unwilling or unable to comply with the protocol
* Pregnant woman or breastfeeding
* Contraindications to treosulfan

  * Hypersensitivity to the active substance
  * Active non-controlled infectious disease
  * Fanconi anaemia and other DNA breakage repair disorders
  * Administration of live vaccine
* Contraindications or any circumstance that precludes the use of the drugs involved in the protocol (especially Thiotepa and Fludarabine)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-01-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Disease and rejection free survival | 12 months after haplo-identical transplantation

SECONDARY OUTCOMES:
Incidence of acute GVHD grade 2/4 | at 100 days
  Acute GVHD will be assessed according to the modified Glucksberg classification
Incidence of acute GVHD grade 3 or 4 | at 100 days
  Acute GVHD will be assessed according to the modified Glucksberg classification
Engraftment | at 100 days
  Engraftment is defined as neutrophil engraftment : neutrophil count at 0.5G/L or higher for more than 3 consecutive days after transplantation, it should be confirmed by a donor chimerism and platelet recovery: platelet engraftment will be defined as first day of platelet > 20G/L without transfusion the last 7 days assessed on day 100
Incidence of chronic GVHD | at 12 months
  Chronic GVHD will be assessed according to the revised Seattle criteria
Non-relapse mortality | at 12 months
Overall survival | at 12 months
Relapse incidence | at 12 months
Rejection incidence | at 12 months
Time to neutrophil engraftment | at 100 days
  Neutrophil engraftment is defined as neutrophil count at 0.5G/L or higher for more than 3 consecutive days after transplantation, it should be confirmed by a donor chimerism
Time to platelet engraftment | at 100 days
  Platelet engraftment is defined as first day of platelet > 20G/L without transfusion the last 7 days assessed on day 100
Infection incidence | at 100 days
Infection incidence | at 12 months
Cytokine profile during transplantation | day-6
Cytokine profile during transplantation | at day 0

IPD SHARING:
Plan to Share IPD: Undecided